CLINICAL TRIAL: NCT02716688
Title: A Phase Ⅱ Study of S-1 With Concurrent Radiotherapy in Elderly Esophageal Cancer Patients
Brief Title: S-1 and Radiotherapy for Elderly Esophageal Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Shiliang Lv, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangPPH02
Record Dates: First submitted 2016-02-11; First posted 2016-03-23 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer; S-1; Radiotherapy
Keywords: Esophageal cancer; Radiotherapy; elder; S-1
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination); Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy and S-1 arm (Experimental): Radiotherapy will be delivered with a daily fraction of 1.8 Gy to a total dose of 50.4 Gy. Preplanned concurrent S-1 (70mg/m²/day) will be administered on Day 1 for 14 days, every 3 weeks. After dCRT, maintenance S-1 will be given up to two cycles.
  Interventions: Drug: S-1; Radiation: radiotherapy

INTERVENTIONS:
Drug: S-1 — S-1 will be administered orally twice daily for 14 days at a dose of 70 mg/m2/day with concurrent radiotherapy for 2 cycles. Patients who showed a response greater than that of stable disease underwent additional S-1 until disease progression, serious adverse events, or patient refusal up to four cycles.
Radiation: radiotherapy — Radiotherapy wiil be delivered with a daily fraction of 1.8 Gy to a total dose of 50.4 Gy.
  Other Names: Irradiation

SUMMARY:
To investigate the efficacy and toxicity of S-1 with concurrent radiotherapy in older patients with esophageal cancer.

DETAILED DESCRIPTION:
Older patients with esophageal cancer have been correlated with poor prognosis because of having little chance to receive aggressive local therapy, including concurrent chemoradiotherapy. In this phase II trial, the efficacy and toxicity of S-1 with concurrent radiotherapy will be investigated in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed esophageal carcinoma;
2. ECOG performance status: 0-1;
3. No treatments prior to enrollment;
4. At least one measurable lesion on CT, MRI or esophageal barium exam;
5. Normal functions of heart, lung, liver, kidney and bone marrow;
6. Blood exams qualified for chemotherapy, which included hemoglobulin ≥9 g/dl, neutrophil ≥1.5×109/L and platelet (PLT) ≥100×109/L, creatinine ≤1.5 UNL;
7. Informed consent signed.

Exclusion Criteria:

1. Prior treatments of chemotherapy or irradiation;
2. Poor bone marrow, liver and kidney functions, which would make chemotherapy intolerable;
3. Contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis;
4. Participating in other clinical trials;
5. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
6. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
response rate | week 4
  Response rate will be done after 4 weeks following the last radiotherapy session.

SECONDARY OUTCOMES:
Progression-free survival | year 0 - year 2
  Progression-free survival (PFS) will be calculated from the date of CCRT initiation to the date of documented failure (local recurrence or metastasis occurrence) or the date of the last follow-up for those remaining.
Acute and late toxicities assessed based on the common toxicity criteria for adverse events version 3.0 (CTCAEv3.0) | year 0 - year 1
  Acute and late toxicities will be assessed based on the common toxicity criteria for adverse events version 3.0 (CTCAEv3.0).
Overall survival | year 0 - year 2
  Overall survival (OS) wiil be determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.

OTHER OUTCOMES:
Dysphagia score | month 0 - month 6
  Dysphagia score was measured according to the following scale: 0, able to consume a normal diet; 1, able to swallow certain solid foods; 2, able to swallow only semisolid foods; 3, able to swallow liquids only; and 4, unable to swallow anything.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China